CLINICAL TRIAL: NCT04051983
Title: iVision - Development of a Game-based Therapy for Children With Cerebral Visual Impairment
Acronym: iVision
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other); KU Leuven (Other); Free University of Brussels (Other); University Ghent (Other); Ganspoel (Unknown)
Responsible Party: Sponsor
Other Study IDs: S61226
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Visual Perceptual Weakness (Disorder); Cerebral Visual Impairment
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the present study is to develop a therapeutic, adaptive, and enjoyable game that will be used by children with CVI between the mental age of 3 and 12 years. Such a game will be easy to use and implement by the children, their parents, and therapists.

DETAILED DESCRIPTION:
The aim of this project is to develop a novel and adaptive gamified visual perceptual therapy platform for children with cerebral visual impairment.

This is a multi-centered study involving multiple partners, namely KU Leuven, VUB, UGent, and a subcontracted game developer. Children and parents will take part during different phases of the research project as described in detail in the different phases below.

Phase I: Quantification of the visual profile (WP1) A quantification of the visual profile of children with CVI will be made by KU Leuven. This will be done using the results conducted at consultations at the CVI clinic at the Centre For Developmental Disabilities Leuven, Centrum Ganspoel, and the CP Reference Centre. A group of 50 children with CVI will be retrospectively recruited and results from their perceptual tests will be used to quantify their visual profile.

Phase II: Definition of user and technical requirements (WP1). A definition of user requirements for the development of the software and mini-games will be identified based on at least two focus groups involving parents and therapists. Two focus groups with parents/caretakes and therapists (one for each age group of the children) each lasting maximum three hours with a limit of 10 participants.

There is also a step involving the technical foundations and development of building blocks, but this will not involve patients, therefore it is not discussed further (WP2).

Phase III: Development and validation of the Relative Enjoyment Scale for Primary School Children (RES-C;WP1). The development and validation of the Relative Enjoyment Scale for Primary School Children (RES-C) instrument will be developed considering not just the affective and the cognitive dimensions of RES-C, but also its socio-cultural embeddedness, by measuring the child's experience in relation to what they have encountered before their experience horizon. The questionnaire will be developed by structured individual interviews with 20 children (10 from each age group).

Phase IV: Initial prototype testing (WP3). During prototype development a game design document will be created, specifying what the core gameplay mechanics are, how the game will look in terms of art and customizable visuals/gameplay. VUB will use the coded visual perceptual profile of the children and map these profiles onto the appropriate game difficulty levels for each child. Prototype testing will occur using structured interviews with 20 children (10 from each age group) while they play the game.

The present study will end in October 2020. Phase I, Phase II, and Phase III will be completed by October 2019. Phase IV will be completed by October 2020.

ELIGIBILITY:
Inclusion Criteria:

* Visual perceptual deficits or diagnosed with CVI
* Gross Motor Function Classification (GMFCS) level I-IV
* Two age groups; 3-7 and 8-12 years of mental age

Exclusion Criteria:

* mental age below 3 and above 12 years of mental age
* severely limited motor abilities (cerebral palsy with a gross motor function classification level V)
* severely limited or unable to express their experiences with the game due to serious speech disorders, deafness, autism
* visual acuity of ≤ 3/10

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fifty children will be recruited from the consultations at the CVI clinic at the Centre For Developmental Disabilities Leuven, from Centrum Ganspoel, and the CP reference Centre of the UZ Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
L94 Visual Perceptual Battery | 25 minutes.
  L94 is an object recognition battery for children aged 3-6 years. The test is composed of 5 computer tasks, [visual matching (VISM), overlapping line drawings (OVERL), line drawings occluded by noise (NOISE), De Vos task (DE VOS), unconventional object views (VIEW). (Ortibus et al., 2009)
Test of Visual Perceptual Skills (TVPS) | 30 minutes.
  TVPS-3 is a standardized and norm-referenced task for children age 4-13 years that uses a response format suitable for all children, including those with disabilities. It includes subtasks of visual discrimination, visual memory, visual-spatial relationships, form constancy, visual sequential memory, figure ground, and visual closure (Martin et al., 2006).
Developmental Test of Visual - Motor Integration (Beery VMI) | 20 minutes.
  Beery a standardized and norm-referenced screening tool for visual-motor deficits. It includes updated norms for ages 2 through 18. The VMI helps assess to what extent children can integrate their visual and motor abilities. In addition to a copying task, the child also performs a visual perception matching task of the same constructs seen before in the copy task, and a motor coordination task, developed to assess the supplementary motor deficits. (Beery et al., 2010).
Developmental Neuropsychological Assessment (NEPSY-II-NL) | Subtests geometric puzzles and arrows, 20 minutes.
  NEPSY-II-NL is a customizable cognitive assessment tool for children aged 5 to 16 years. It assesses six domains with one integrated instrument, composed of different normed subtests. Among those, visual attention and visuospatial functions, are routinely performed in the diagnostic work up of children with (a suspicion of) CVI. (Korkman, 1998).
Revisie Amsterdamse Kinderintelligentie Test (RAKIT) | Subtests Hidden figures and Figure recogntion, 20 minutes.
  RAKIT is a paediatric intelligence test, with reference values from a Dutch population of children 4-12.5 years of age. From this test, the subtest "Vertelplaat" is used to evaluate the ability to tell a logic story from a crowded scene, thereby evaluating object recognition, figure ground perception and scene perception (Bleichroth et al., 1987).
Relative Enjoyment Scale for Primary School Children adapted for cerebral visual impairment (RESC-CVI) | 10 minutes
  The RES-C measures enjoyment by relating it subjectively to a series of other activities which are part of the 'experience horizon' of a child using visual analogue scales (Van Looy et al., 2016)
Preschool judgment of line orientation (PJLO) | 10 minutes.
  The PJLO is an extension of the Benton judgment of line orientation task and is administered to children between the age of 3.25 and 6 years. This test includes 24 items where the orientation of one or two target lines needs to be matched to 2, 4, or 11 choices (Stiers et al., 2005).
Motion perception tasks | 20 minutes.
  Motion perception tasks measure motion-defined form, global motion coherence, motion speed, and biological motion, and can be administered to children between the age of 4 and 6 years. In motion-defined form, an object is concealed in a random dot kinematogram and the child is required to identify the image seen. In global motion coherence, the child indicates in which half of the display, left or right, a coherently moving strip forming a horizontal bar is located. In motion speed, two contours of a car are shown next to each other with moving dots inside, and the child indicates in which car the dots are moving at the highest speed. In biological motion, two dot matrices are shown, one is a human-point light walker (walking man) and the other one is a phasescrambled point-light figure, and the child should indicate the walking man (Van der Zee et al., 2019).
The Flemish cerebral visual impairment questionnaire (FCVIQ) | 10 minutes.
  The FCVIQ is a 46-item screening tool for CVI filled out by caregivers using a binary response format (yes or no). This tool screens for visual perceptual difficulties in daily life (Ortibus et al., 2011).

SECONDARY OUTCOMES:
Snijders-Oomen Non-verbal intelligence test (SON-R 6-40) | 60 minutes.
  The SON-R 6-40 consists of four subtests containing two or three parallel series of twelve to thirteen items with increasing difficulty. The testing procedure of this test is adaptive, whereby the starting point of a series is decided on basis of the score on the previous series of the subtest.
Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III-NL) | Non-verbal subtests, 45 minutes.
  Third Edition (WPPSI-III) is designed to test intelligence (cognitive ability) in children ages 2 years 6 months to 7 years 3 months. The test consists of 14 subtests from which five subtests measure the non-verbal intelligence.

CONTACTS AND LOCATIONS:
Overall Officials: Els Ortibus, Professor, Study Director — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-brabant, Belgium

IPD SHARING:
Plan to Share IPD: No